CLINICAL TRIAL: NCT00307411
Title: Effects of Growth Hormone on Body Fat Distribution, Insulin Action and Cardiovascular Risk Factors in Middle-Aged Men With Metabolic Syndrome
Brief Title: Effect of Growth Hormone in Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUHK 4470/05M
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-04-04 (Estimated); Status verified 2006-03

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Growth Hormone

INTERVENTIONS:
Drug: Growth hormone

SUMMARY:
Investigating the effect of low dose growth hormone therapy on body fat composition, insulin sensitivity and metabolic profiles in middle-aged men with metabolic syndrome and low insulin-like growth factor (IGF-1) level.

DETAILED DESCRIPTION:
Metabolic syndrome, a constellation of glucose intolerance, hypertension, dyslipidemia, obesity, pro-inflammatory and prothrombotic state culminating to development of premature cardiovascular diseases is a serious public health problem with significant impact on life expectancy, societal productivity and quality of life of those afflicted with it. Insulin resistance has been proposed as the key linking factor for the metabolic syndrome. Although the underlying mechanism for the development of insulin resistance, diabetes and metabolic syndrome is not fully understood, increasing evidence suggests that neurohormonal dysregulation plays a pivotal role in causing this growing health hazard. In our previous study of 307 middle-aged men, low insulin-like growth factor (IGF)-1 level was independently associated with insulin resistance and metabolic syndrome, especially amongst those with positive family history of diabetes. Replacement with growth hormone has been shown by other researchers to reduce body fat and improve metabolic profiles in patients with adult growth hormone deficiency and type 2 diabetes.

We hypothesize that treatment with growth hormone can lead to reduction of body fat, insulin resistance and cardiovascular risk factors in men with metabolic syndrome. This will be a 12-month prospective, randomized, double-blind, placebo-controlled study using growth hormone treatment in middle-aged men with metabolic syndrome. The primary outcome measure will be body fat distribution, including changes in visceral and mesenteric fat, whereas secondary outcome measure will be insulin sensitivity, and tertiary outcome will be variable parameters of metabolic syndrome.

The results of this study will have important impact on the treatment of patients with metabolic syndrome, and our understanding of the role of growth hormone in the pathogenesis of insulin resistance, diabetes and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 50 Chinese men
* Metabolic syndrome as defined according to 1998 World Health Organisation with modification using Asian definition for obesity (body mass index 25kg/m2, waist circumference 80cm in women and 90 cm in men)
* Low IGF-1 level or IGF-1 level in low normal range (<200 ug/L)

Exclusion Criteria:

* Any malignancy within the past 5 years
* A diagnosis of acromegaly
* Uncontrolled hypertension (systolic blood pressure >180mmHg or diastolic blood pressure>105mmHg)
* A history of carpel tunnel syndrome
* Poor glycemic control (HbA1c>8%)
* Diabetic microangiopathy
* Previous cardiovascular event
* Anaemia as defined as haemoglobin <11g/dL
* Active thyroid diseases
* Any medical illness that will render the subject vulnerable to fluid retention state, e.g. renal impairment, heart failure or as judged by the investigators as ineligible to participate the study.

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-08; Study Completion 2007-07

PRIMARY OUTCOMES:
Change in percentage of body fat from baseline.

SECONDARY OUTCOMES:
Examine the percentage change from baseline in insulin sensitivity, various indices of metabolic syndrome of growth hormone treatment will be compared to placebo arm.

CONTACTS AND LOCATIONS:
Overall Officials: Alice PS Kong, M.B.,Ch.B., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong SAR, China